CLINICAL TRIAL: NCT02225483
Title: Phenotypic Heterogeneity in Hemophilia A: An Investigation of the Role of Platelet Function
Status: Completed | Type: Observational
Sponsor: CancerCare Manitoba (Other)
Collaborators: The Hospital for Sick Children (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: H2013:304
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemophilia A: Boys with Factor VIII coagulant activity less than or equal to 1%.

SUMMARY:
The is study will examine whether variation in clinical bleeding frequency and severity among boys with severe Hemophilia A (Factor VIII deficiency) is associated with variations in laboratory measurements of platelet activity.

ELIGIBILITY:
Inclusion Criteria:

* documented circulating FVIII level of ≤1%
* age 3 - 20 years
* may be on primary or secondary prophylaxis
* granting of informed consent

Exclusion Criteria:

* measurable inhibitor level at the time of enrollment
* ingestion of aspirin/supplement known to influence platelet function within 14 days of blood sampling, or ibuprofen within 3 days

Ages: 3 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys with severe Hemophilia A, Factor VIII coagulant activity less than or equal to 1%
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Procoagulant platelet-derived microparticle formation | At time of enrollment
Platelet aggregation | At time of enrollment
  Whole blood platelet aggregation responses

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Hospital for Sick Children, Toronto, Ontario